CLINICAL TRIAL: NCT01479049
Title: The Myocardial Protective Effects of a Moderate-potassium Blood Cardioplegia in Pediatric Cardiac Surgery：a Randomized Controlled Trial
Brief Title: The Myocardial Protective Effects of a Moderate-potassium Blood Cardioplegia in Pediatric Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XJXZ2009-1010
Record Dates: First submitted 2011-10-07; First posted 2011-11-24 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Congenital Heart Disease
Keywords: congenital heart disease; cardiac surgery; cardiopulmonary bypass; cardioplegia
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MP group (Experimental): Hearts are arrested with cold blood cardioplegia with moderate potassium concentration (K+, 10mmol/L) during cardiac surgery.
  Interventions: Drug: MP (moderate potassium) group
- HP group (Active Comparator): Hearts were arrested with cold blood cardioplegia with high potassium concentration (K+, 20mmol/L) during cardiac operation
  Interventions: Drug: HP (High potassium) group

INTERVENTIONS:
Drug: MP (moderate potassium) group — Hearts were arrested with cold blood cardioplegia with moderate potassium concentration (K+, 10mmol/L)during cardiac operation
  Other Names: moderate potassium cardioplegia
  Arms: MP group
Drug: HP (High potassium) group — Hearts are arrested with cold blood cardioplegia with high potassium concentration (K+, 20mmol/L)during cardiac operation.
  Other Names: High potassium cardioplegia
  Arms: HP group

SUMMARY:
The investigators previously investigated the cardioprotective effect of an adenosine-lidocaine cardioplegia with moderate-potassium (K+, 10.0 mmol/L) in pediatric cardiac surgery, which was associated with better myocardial protective effects when compared with conventional high-potassium cardioplegia. However, this cardioplegia could not be sucked back into the cardiopulmonary bypass (CPB) circuit because of excessive hemodilution and severe systemic hypotension induced by adenosine. Therefore, the investigators supposed that a moderate-potassium (K+, 10.0 mmol/L) blood cardioplegia without adenosine could also arrest the heart and have better myocardial protective effects compared with conventional hyperkalamic cold blood cardioplegia during cardiac operations without excessive hemodilution and systemic hypotension.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients (body weight<10 kg)
* congenital heart diseases and scheduled for a repair operation with CPB in the Department of Cardiovascular Surgery, Xijing Hospital.

Exclusion Criteria:

* other systemic diseases

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2009-10; Primary Completion 2010-03 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
post-operative Serum cTnI concentration decreased significantly in 24hours | 24h after myocardial reperfusion
  myocardial injury could be sensitively reflected by post operative Serum cTnI concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenxiao Jin, PhD, Principal Investigator — Department of Cardiovascular Surgery, Xijing Hospital
Locations (1):
- Department of Cardiovascular Surgery, Xijing Hospital, Xi'an, Shaanxi, China